CLINICAL TRIAL: NCT07314307
Title: Vaccine Effectiveness of One Dose of the Nonavalent Human Papillomavirus (HPV) Vaccine Among Young-adult Women in Sweden Among Women Participating in a Clinical Trial of Concomitant HPV Vaccination and Screening
Acronym: FASTER1DOSE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Joakim Dillner, Professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-07145
Record Dates: First submitted 2025-09-10; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-09

CONDITIONS: Incident HPV16, 18, 31, 33, 45, 52 or 58 Infection
Keywords: HPV; Vaccine effectiveness; one dose; Even Faster
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine nonavalent; Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Concomitant HPV vaccination and screening intervention arm (Experimental): Eligible women were invited by letter, push notification (via their personal mobile telephones) to attend a vaccination site for concomitant HPV vaccination (with the nonavalent vaccine Gardasil 9) and HPV-based cervical screening (using a self-sample). After 3 years women who had received their first vaccine dose were invited to receive a second dose of the nonavalent HPV vaccine and to give a second screening sample.
  Interventions: Biological: Gardasil 9 2 dose regimen
- Unvaccinated comparison group (No Intervention): The unvaccinated comparison group will be comprised of unvaccinated women attending routine screening in Sweden (whole trial or Stockholm region in the piloting phase).

INTERVENTIONS:
Biological: Gardasil 9 2 dose regimen — Women ages 22-26 will be offered concomitant vaccination (1 dose of Gardasil9) and HPV screening. A second dose of Gardasil9 will be administered 3 years later.
  Arms: Concomitant HPV vaccination and screening intervention arm

SUMMARY:
This study aims to evaluate the vaccine effectiveness of 1 dose the nonavalent human papillomavirus (HPV) vaccine against HPV16, 18, 31, 33, 45, 52, and 58 infection among young adult women in Sweden participating in a nationwide HPV elimination trial.

DETAILED DESCRIPTION:
HPV vaccination is the 1st pillar in the World Health Organization's (WHO) strategy to eliminate cervical cancer as public health problem, defined as an incidence of under 4 per 100,000 women-years globally. Licensed prophylactic HPV vaccines are highly efficacious in preventing HPV infection and associated cancers. At the time of licensure, the first-generation vaccines were licensed with a 3-dose schedule, and subsequently with a 2-dose schedule for women aged 15 and under. However, based on promising findings from observational studies of high vaccine effectiveness after only one dose, and subsequent clinical trials, the Strategic Advisory Group of Experts on Immunization (SAGE) recommended an off-label HPV vaccination regimen of one dose for girls and women from the age of 9 to 20 years-old. However, for women aged 21 or older a 2-dose schedule is still recommended by the WHO.

This nationwide trial of concomitant HPV vaccination among women aged 22 to 30-years-old in Sweden is a unique opportunity to evaluate the vaccine effectiveness of one dose of HPV vaccination among women over the age of 20 years old. Studies on the efficacy and effectiveness of one dose among women over the age of 20 years old are scarce and of varying quality. The findings of this study will be crucial to inform public health decision makers and in contributing to the evidence base for assessing if the 2-dose schedule recommendation among women over 20-years-old is still warranted.

ELIGIBILITY:
Inclusion Criteria:

* Eligible women will include resident women born between 1994-1999 (1993-1999 in the non intervention arm), who have not opted out of the screening program and who consent to participate in the study.

Exclusion Criteria:

* Known history of severe allergic reaction or hypersensitivity to any of the components of the HPV vaccine.For GARDASIL 9: Amorphous aluminium hydroxyphosphate sulphate adjuvant, Sodium chloride, L-histidine, Polysorbate 80 or Sodium borate
* Known history of immune-related disorders
* Current acute severe febrile illness, except for minor infections such as a cold, mild upper respiratory infection or low-grade fever.
* Administration of immunoglobulin or blood-derived products within 6 months prior to scheduled HPV vaccine first dose
* Current pregnancy (reported)
* Women with a total hysterectomy

Ages: 22 Years to 31 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gender eligibility is based on the sex coded in the personal identification number used in civil society in Sweden.
Enrollment: 150000 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
HPV16, 18, 31, 33, 45, 51, 52, and 58 incident HPV infection | 6 years
  Incidence rate of incident HPV16, 18, 31, 33, 45, 52 or 58 infection 3 years after receiving one dose of the nonavalent vaccine, among the 1994-1999 born women participating in the elimination trial nationwide at the time who were HPV negative at baseline (negative for the specific HPV type in the analysis).

SECONDARY OUTCOMES:
HPV16, 18, 31, 33, 45, 51, 52, and 58 incident HPV infection | 6 years
  Incidence rate of incident HPV16, 18, 31, 33, 45, 52 or 58 infection 3 years after receiving one dose of the nonavalent vaccine, among the 1994-1999 born women participating in the elimination trial in the Stockholm region (the piloting phase), who were HPV negative at baseline (negative for the specific HPV type in the analysis).
HPV16, 18, 31, 33, 45, 51, 52, and 58 incident HPV infection | 6 years
  Incidence rate of incident HPV16, 18, 31, 33, 45, 52 or 58 infection 3 years after receiving one dose of the nonavalent vaccine, among the 1994-1999 born women participating in the elimination trial nationwide at the time who were HPV negative at baseline (negative for the specific HPV type in the analysis) in relation to their previous HPV vaccination history.

CONTACTS AND LOCATIONS:
Overall Officials: Joakim Dillner, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Documents related to the study can be shared. Data, once collected, will be made available.
Supporting Information: Study Protocol, SAP
Time Frame: The study protocol and statistical analysis plan are available.
Access Criteria: Data can be shared with other researchers upon written request.

REFERENCES:
- [Background] Arroyo Muhr LS, Gini A, Yilmaz E, Hassan SS, Lagheden C, Hultin E, Garcia Serrano A, Ure AE, Andersson H, Merino R, Elfstrom KM, Baussano I, Dillner J. Concomitant human papillomavirus (HPV) vaccination and screening for elimination of HPV and cervical cancer. Nat Commun. 2024 May 1;15(1):3679. doi: 10.1038/s41467-024-47909-x. PMID 38693149

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT07314307/Prot_SAP_000.pdf